CLINICAL TRIAL: NCT02156232
Title: Embolization of Large Spontaneous Portosystemic Shunts for the Prevention of Post-TIPS Hepatic Encephalopathy: a Prospective、Open-labeled、Randomized、Controlled Trial
Brief Title: Embolization of Large Spontaneous Portosystemic Shunts for the Prevention of Post-TIPS Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, M.D., Ph.D., Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TIPS-SPSS
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Liver Cirrhosis
Keywords: hepatic encephalopathy (HE); vericeal bleeding; spontaneous portosystemic shunts (SPSS); transjugular intrahepatic portosystemic shunt (TIPS); embolization
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIPS, SPSS Emboliaztion (Active Comparator): The covered stents wil be used for TIPS The SPSS will be embolized during the procedure of TIPS
  Interventions: Procedure: TIPS; Procedure: SPSS embolization
- TIPS alone (Active Comparator): The covered stents will be used for TIPS No embolization of SPSS will be performed during TIPS
  Interventions: Procedure: TIPS

INTERVENTIONS:
Procedure: TIPS — TIPS is performed with a standard technique. TIPS revision will be planned if any evidence of shunt dysfunction is observed.
Procedure: SPSS embolization — Embolization of SPSS will be conducted via the same jugular vein before TIPS implantation. The major procedures included (a) angiography of SPSS after successful intrahepatic puncture of a branch of the portal vein and (b) embolization of SPSS with coils of varying diameters or Amplatzer Vascular Plug, which resulted in the SPSS disappearing at postembolization angiography.
  Arms: TIPS, SPSS Emboliaztion

SUMMARY:
The purpose of this study is to determine whether transjugular intrahepatic portosystemic shunt (TIPS) combined with large spontaneous portosystemic shunts embolization are effective in the prevention of hepatic encephalopathy (HE).

DETAILED DESCRIPTION:
Transjugular intrahepatic portosystemic shunt (TIPS) has been used for more than 20 years since 1988 to treat some of the complications of portal hypertension, especially variceal bleeding and ascites refractory to conventional therapy. However, this procedure has two major disadvantages: shunt dysfunction and hepatic encephalopathy (HE). Notabley, the use of expanded polytetrafluoroethylene (ePTFE)-covered stent has significantly reduced the risk of shunt dysfunction, but the post-TIPS HE remains a problem even with these new stents.

The incidence of post-TIPS HE ranges between 5% and 35% HE during the first year and tends to be particularly frequent during the first months after TIPS and less common with time. Meta-analysis has that increased age, prior HE and higher Child-Pugh class/score were the most robust predictors for post-TIPS HE.

There is no consensus on the management of post-TIPS HE. Episodic HE after TIPS can be treated traditionally. The cornerstones of the treatment of this type of HE are the identification and treatment of the precipitating event and the general support of the patients. Refractory HE not responding to standard treatment is, in our opinion, the most important problem faced when a patients has to be treated with TIPS. In some cases, the occurrence of this complication may deeply reduce the patient's quality of life and the cure may be worse than the disease. Refractory HE can be treated by reducing the diameter of the stent or by occluding the shunt. However, the procedure is not without dangers and may not solve the problem in all patients, and the complications of portal hypertension, such as varices or refractory ascites, which were supposed to be managed by the TIPS, may recur as a consequence of shunt reduction or occlusion.

Besides, there are no established methods or drugs to effectively prevent the occurrence of HE after TIPS. One possibility is the use of stents with a small diameter, since post-TIPS HE was related to the amount of blood shunted. Riggio et al. compared the incidence of HE after TIPS created with 8-or 10-mm PTFE-covered stents and the study was stopped because of higher complications due to portal hypertension after TIPS in the 8-mm group. Our center performed a RCT to evaluate the effectiveness of L-ornithine-L-aspartate (LOLA) on plasma ammonia in cirrhotic patients after TIPS. Another RCT reevaluateing the effect of TIPS with 8- or 10-mm covered stent for the prevention of variceal rebleeding in cirrhotic patients was also undergoing.

But for those with large spontaneous portosystemic shunts(SPSS), embolization might also represent a therapeutic target.SPSS is, as the name implies, potential communications between the portal venous circulation and the systemic venous circulation that can open, develop, and potentially grow to enable flow within them when one of these circulations (portal or venous) has high pressure or is obstructed or both in an effort to reduce pressure or bypass an obstruction or both. SPSS mainly include splenorenal shunt, gastrorenal shunt, paraesophageal vein, paraumbilical vein, et al. For patients with decompensated cirrhosis, the portal vein pressure increased significantly and some blood were diverted to the systemic circulation by collateral vessels between the splenorenal vein, short gastric veins, posterior gastric vein, and so on, namely SPSS. The nature history of SPSS in patients with liver cirrhosis is still unclear. Most patients were diagnosed by chance.

Previous reports have suggested that the incidence of SPSS was 16% in patients with liver cirrhosis and portal hypertension and the incidence of refractory HE was about 46%. A study published in 2005 revealed that about 71% of the patients with cirrhosis with refractory HE have large SPSS. Therefore, the presence of a SPSS not only provides an explanation for the persistence or recurrence of HE despite an acceptable liver function, it might also represent a therapeutic target. Nowadays, several series have reported embolization of large SPSSs for the treatment of chronic therapy-refractory HE.To date, no data was about the safety and efficacy of embolization of large SPSS in the prevention of post-TIPS HE.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Dignosis of liver cirrhosis (clinical or by liver biopsy)
* Admission due to variceal bleeding occurred 5 to 42 days prior and standard treatment for secondary prophylaxis failed
* Confirmed spontaneous portosystemic shunts in abdominal imagings
* Sum of targeted spontaneous portosystemic shunts diameters greater than half the diameter of portal vein

Exclusion Criteria:

* Hepatic carcinoma and/or other malignancy diseases
* Portal vein thrombosis (≥50% of the lumen)
* Budd-Chiari syndrome
* Child-Pugh score>13 points
* Sepsis
* Spontaneous bacterial peritonitis
* Uncontrollable hypertension
* Serious cardiac or pulmonary dysfunction
* Renal failure
* With TIPS contraindications
* Spontaneous recurrent hepatic encephalopathy
* Previous TIPS or collateral embolization
* Pregnancy or breast-feeding
* History of liver transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-06-15; Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Number and severiy of participants with overt hepatic encephalopathy | 2 years

SECONDARY OUTCOMES:
Number of participants with variceal rebleeding | 2 years
Number of participants with shunt dysfunction | 2 years
Change of liver function | 2 years
All-cause mortality | 2 years
Adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, PhD,MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China